CLINICAL TRIAL: NCT03460561
Title: Peri-operative Rectus Sheath Fentanyl-Levo Bupivacaine Infusion Versus Thoracic Epidural Fentanyl-Levo Bupivacaine Infusion in Patients Undergoing Major Abdominal Cancer Surgeries With Medline Incision
Brief Title: Peri-operative Rectus Sheath Block Versus TEA Abdominal Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, Principal Investigator, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: South Egypt Cancer Institute
Record Dates: First submitted 2018-02-21; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Abdominal Cancer
Keywords: TEA; Rectus sheath block; Major abdominal cancer surgery
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEA group (Active Comparator): peri operative thoracic epidural block (TEA) via fentanyl-levo bupivacaine infusion.
  Interventions: Procedure: Thoracic epidural block (TEA)
- RSB group (Active Comparator): peri operative rectus sheath block (RSB) via fentanyl-levo bupivacaine infusion.
  Interventions: Procedure: Rectus sheath block (RSB)

INTERVENTIONS:
Procedure: Thoracic epidural block (TEA) — Under complete aseptic precautions and before induction of GA, thoracic epidural catheter was inserted using a 17 gauge, Tuohy epidural needle by a midline approach. T9-T10 interspace was chosen for the injection after skin infiltration by 5 mL of lidocaine 1%. The epidural space was identified by the loss of resistance technique then the catheter was introduced 2 cm into the epidural space, and epidural test dose of 3 mL of lidocaine 2% with 1:200,000 adrenaline was injected to exclude vascular or subarachnoid position.
  Other Names: Thoracic epidural analgesia
  Arms: TEA group
Procedure: Rectus sheath block (RSB) — Under aseptic technique, the rectus muscle was imaged with the ultrasound probe, A broadband (5-12 MHz) linear array probe of Sonosite ™ 3000 ultrasound (FUJIFILM, Sonosite EDGE II -UAS) in a transverse orientation at or immediately above the level of the umbilicus, with an imaging depth of 4-6 cm.
  Inserting the needle: An 18G Tuohy needle was introduced few millimeters from the probe using an in plane technique in an angle of 45 degrees to the skin. (posterior rectus sheath and fascia transversalis). Under direct vision, the needle tip was advanced to the desired position where 20 mL of (levo-bupivacaine 0.25% Fentanyl 30 μg) were injected causing hydro dissection of the rectus muscle away from the posterior rectus sheath. The technique is repeated on the opposite side.
  Arms: RSB group

SUMMARY:
Thoracic epidural analgesia (TEA) can be considered the gold standard for postoperative analgesia in major abdominal surgeries, as proved by a lot of number of systematic reviews and meta-analyses have demonstrated that TEA was associated with superior postoperative analgesia, better patients' outcomes, reducing (systemic opiate requirements, ileus and pulmonary complications).

The rectus sheath block (RSB) is effective for the surgeries that necessitated midline abdominal incisions as local anesthetics instillation will be within the posterior rectus sheath bilaterally providing intense analgesia for the middle anterior wall from the xiphoid process to the symphysis pubis in adults.

DETAILED DESCRIPTION:
The aim of the study was to assess the efficacy and safety of intra and post operative ultrasound-guided RSB versus intra and post operative TEA and to investigate role of Fentanyl as an adjuvant in both RSB and TEA, in patients undergoing elective major abdominal surgery with midline abdominal incisions.

Pre operative medications in the form of oral ranitidine tablet, 50 mg and lorazepam tablet, 3 mg on the night of surgery were given to all patients.

All patients were taught- The day before surgery- how to evaluate their own pain intensity using the visual analog scale (VAS), scored from 0 to 10 (where 0=no pain and 10= worst pain imaginable) and how to use the patient controlled analgesia (PCA) device (Abbott Laboratories, North Chicago, IL, USA).

Patients were randomly assigned into two groups, 50 patients each, by using opaque sealed envelopes containing a computer generated randomization schedule; the opaque envelopes were sequentially numbered and were opened before application of anesthetic plan.

TEA group (No. =50); where patients received TEA in conjunction with GA, intraoperative analgesia was started before skin incision by epidural bolus dose of 0.1 ml ∕ kg of 0.125% levo-bupivacaine ∕ fentanyl 2 µg ∕ ml. Postoperative analgesia was provided through Patient controlled epidural analgesia (PCEA) for 48 hours postoperative, by continuous infusion of a mixture of (0.0625% levo-bupivacaine ∕ fentanyl 2 µg ∕ ml) in a dose of of 0.1 ml ∕ kg, and bolus dose of 3 ml, lockout interval of 20 minutes).

RSB group (No. =50); combined general plus US guided rectus sheath block (group-RSB): where 20 mL of (0.25% levo-bupivacaine + fentanyl 30 µg) in saline were injected into the rectus sheath plane on either side under direct US visualization 15 minutes before skin incision.

And before closure of abdominal wall, bilateral surgically placed catheters in rectus sheath plane for post operative analgesia for 48 hours.

Postoperative analgesia was as following; injection of 20 mL of (0.125% levo-bupivicaine +Fentanyl 30 μg) every 12 hours in to each catheter, A postoperative rescue analgesia with intravenous Fentanyl per a titration protocol (Fentanyl 30 μg IV as a bolus dose that could be repeated every 10 minute) was employed if visual analog pain scale (VAS) ≥4.

ELIGIBILITY:
Inclusion Criteria:

* 100 adult patients, classified as American Society of Anesthesiologists (ASA) grade II and III, scheduled for elective major abdominal cancer surgery were consecutively enrolled.

Exclusion Criteria:

* We excluded from the study; patients who refused the study, Patients with coagulopathy, active neurological disease, cutaneous disorders at the epidural insertion site, and who were allergic to the studied medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
assessing a change in VAS score with cough | at 0, 4, 8, 12, 18, 24, 36 and 48 hours post operative.
  assessing a change in Pain severity by VAS score with cough (0-10) 0=no pain 10=worst pain ever

SECONDARY OUTCOMES:
assessing a change of MAP | at baseline , 4, 8, 12, 18, 24, 36 and 48 hours post operative.
  assessing a change in Mean arterial pressure from baseline reading

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A. Elzohry, MD, Principal Investigator — Principal Investigator
Locations (1):
- South Egypt Cancer Institute, Assiut University, Arab Republic of Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided